CLINICAL TRIAL: NCT02159742
Title: Prospective Follow-up of Outcomes in Patients Receiving Photodynamic Therapy for Neoplastic Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 06911
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Neoplastic Disease
Keywords: Adult subjects; history; treatment; photodynamic therapy
MeSH Terms: conditions — Neoplasms | interventions — Data Collection; Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cohort 1
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection
  Other Names: Prospective/retrospective data will be collected from medical records of patients who have received PDT for; neoplastic diseases.

SUMMARY:
From 1996-present, we have used photodynamic therapy (PDT) to treat a number of neoplastic diseases both on prospective research protocols (for head and neck cancer, pleural malignancies, peritoneal carcinomatosis or sarcomatosis and prostate cancer) as well as for FDA approved and off label or compassionate exemption indications (neoplasms of the skin, bronchus, esophagus, head and neck and pleura). The goal of this treatment is to maximize quality of life and organ function while minimizing the chance of tumor recurrence. As such, we would like to retrospectively review the treatment parameters of all patients who undergo/underwent PDT (including operative notes and photodynamic therapy records) and treatment outcomes (including all organ functions, performance status, tumor recurrence, laboratory values and any other data present in the routinely documented follow up visits). For patients who have died or were lost to follow-up prior to initiation of this study, a retrospective review of available data will be performed. For patients who are still being actively followed after PDT or who receive PDT after the initiation of this study, informed consent will be obtained for obtaining continued follow-up data prospectively and any previous data will be collected retrospectively.. These subjects will continue to receive care from their current physicians according to standard medical practice and no attempt will be made to alter the types of follow-up, radiologic or other diagnostic studies or medical treatment as a result of enrollment in this study. All data will be de-identified and added to our already existing PDT treatment outcome databases for outcomes analysis, quality improvement and reporting of results in abstract and manuscript forms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be age 18 or greater
* Subjects will have undergone PDT for a diagnosis of neoplastic disease under the direction of a Penn physician.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective/retrospective data will be collected from medical records of patients who have received PDT for neoplastic diseases.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Survival and disease free | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Keith Cengel, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States